CLINICAL TRIAL: NCT02876094
Title: A Pilot, Open-Label, Dose Response Study Investigating the Effect of Low-Dose Celecoxib on SMN2 in Patients With Spinal Muscular Atrophy (SMA)
Brief Title: Effect of Low-Dose Celecoxib on SMN2 in Patients With Spinal Muscular Atrophy
Acronym: SMA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention
Sponsor: Hugh McMillan (Other)
Collaborators: Families of Spinal Muscular Atrophy (Other); Gwendolyn Strong Foundation (Other)
Responsible Party: Sponsor-Investigator, Hugh McMillan, MD, MSc, FRCPC, FAAN, Pediatric Neurologist, Children's Hospital of Eastern Ontario
Organization: Children's Hospital of Eastern Ontario (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15/22E
Record Dates: First submitted 2016-08-09; First posted 2016-08-23 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Spinal Muscular Atrophy (SMA)
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-label (Experimental): All patients will be treated at each dose of oral once daily celecoxib (40, 80 and 160 mcg/kg) for a period of two weeks, for a total of 6 weeks (42 days) of treatment.
  Interventions: Drug: celecoxib

INTERVENTIONS:
Drug: celecoxib — dose-response
  Other Names: CeleBREX

SUMMARY:
Several factors make the use of celecoxib in human SMA patients appealing including: 1) low-dosing required for potential therapeutic effect (the corresponding dose in humans is much lower than that commonly used in adults and children with; 2) favourable side effect profile of this drug (particularly at the dosing required); 3) the fact that celecoxib crosses the blood brain barrier and 4) demonstration of efficacy in a genetically and pathophysiologically faithful animal mode. The investigators therefore believe that celecoxib is a promising disease modifying therapy for SMA.

DETAILED DESCRIPTION:
This is a pilot, open-label, dose-response study in patients with SMA type II or III. All patients will be treated at each dose of once daily celecoxib (40, 80 and 160 mcg/kg) for a period of two weeks, for a total of 6 weeks (42 days) of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed genetic diagnosis consistent with SMA that can include: SMN1 gene deletions, rearrangements and/or mutations
2. Sufficient clinical information enabling the patient to be classified as either SMA type II or III. (Patients with SMA type II are defined as having achieved the motor milestone of sitting independently for > 30 seconds but not having been able to stand or walk unsupported. Patients with SMA type III are defined as having achieved the motor milestone of standing or walking independently).
3. Confirmed genetic test result indicating number of SMN2 gene copies
4. Age > 2.0 years old at screening
5. Patients weighing at least 12 kg at screening
6. Stable dosing (for at least 3 months) of medications that may affect function of muscle, nerve and/or neuromuscular transmission or gene expression (including but not limited to: coenzyme Q10, creatine monohydrate, nutritional supplements, oral salbutamol, valproic acid, sodium phenylbutyrate, hydroxyurea)
7. Written informed consent obtained from patient and/or parents or legal guardians

Exclusion Criteria:

1. Clinical presentation and/or genetic testing that is not consistent with SMA type II or III
2. Inability or unwillingness to swallow celecoxib suspension
3. Major surgery (scoliosis repair, G-tube insertion) within past 3 months
4. Known hypersensitivity or allergy to celecoxib (including asthma, urticaria and/or other allergic symptoms resulting from prior celecoxib ingestion) or its excipients, or other NSAIDs (non-steroidal anti-inflammatory drugs) including ASA (Acetylsalicylic Acid)
5. Known hypersensitivity or allergy to Ora-Blend® or its excipients
6. Demonstrated allergic-type reaction to sulfonamides
7. Celecoxib use within 2 weeks prior to screening visit
8. Known cardiac (ie. uncontrolled heart failure, cerebrovascular bleeding, hypertension requiring the use of anti-hypertensive medication), hepatic (i.e. severe liver impairment or active liver disease), gastrointestinal (i.e. inflammatory bowel disease; active gastric/duodenal/peptic ulcer disease; or active gastrointestinal bleeding), hematologic (ie. thrombocytopenia defined as platelets < 50,000 or hemophilia), respiratory or renal disease(i.e. severe renal impairment defined as creatinine clearance < 30 mL/min) wherein the use of NSAIDs is contraindicated as per Product Monograph dated 03 March 2015.
9. Concurrent use of medication contraindicated with Celecoxib use (including but not limited to, warfarin, fluconazole, lithium, hydrochlorothiazide)
10. Female who is pregnant or breast feeding
11. Female of child-bearing potential who is sexually active and unwilling or unable to use at least one form of highly effective and one effective method of birth control.
12. Patients participating in any pharmaceutical clinical trial (with active agent) that could impact with the results of this study
13. Inability or refusal to provide informed consent

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
low-dose oral celecoxib administered to patients with SMA type II and III is associated with an increase in the levels of peripheral leukocyte SMN protein compared to baseline | baseline
  1) Investigate change in peripheral leukocyte SMN protein levels from baseline at each dose (40 mcg/kg, 80 mcg/kg, and 160 mcg/kg) of celecoxib.

SECONDARY OUTCOMES:
Safety Profile Measured by Adverse Event Frequency,Type and Severity | 4 weeks post
  1) Determine safety profile as measured by number, type and severity of adverse events reported following administration of low dose celecoxib in patients with type II and III SMA
Recruitment Plan Measured by Number of Potentially Eligible Subjects | 4 weeks post
  Assess understanding of recruitment barriers measured by the number of potentially eligible subjects and response to study recruitment phase.
Compliance Measured by Reported Protocol Deviations | 4 weeks post
  Assess adherence to treatment protocol measured by number of reported protocol deviations.
Eligibility Measured by Number of Screen Failures | 4 weeks post
  Assess appropriateness of eligibility criteria based on number of screen failures.
Delivery Time of Shipped Samples Assessed by Viability | 4 weeks post
  Assess feasibility of shipping laboratory samples to outside centre for analysis. This will be reported based on the time to deliver and the resulting viability of the received samples by either pre or post testing or both if appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Hugh McMillan, MD, Principal Investigator — Children's Hospital of Eastern Ontario Research Institute
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Results will be submitted for presentation at an international meeting and subsequently submitted for publication in a major international peer-reviewed medical journal.